CLINICAL TRIAL: NCT02842346
Title: Correlation Between Umbilical Resistance Index and Fetal Growth: a Pilot Study
Brief Title: Correlation Between Umbilical Resistance Index and Fetal Growth
Status: Completed | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Mehdi Kehila, Dr, University Tunis El Manar
Other Study IDs: CMNTIR
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Umbilical Doppler
Keywords: Ultrasound; umbilical Doppler; resistance index; fetal growth
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: ultrasonography

SUMMARY:
The aim of our study was to investigate the correlation between the umbilical resistance index and weight gain during the third trimester of low-risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant patient with a normally progressing pregnancy and reporting for a prenatal screening ultrasound between 31 and 34 weeks amenorrhea.

Exclusion Criteria:

* -The lack of an ultrasound carried out during the first trimester to confirm the term of the pregnancy.
* A medical condition in the mother: diabetes, high blood pressure or a known chronic illness.
* A medical condition in the fetus: suspicion of fetal hypotrophy (fetal biometrics lower than the 10th percentile), a birth defect (a chromosomal abnormality) during the pregnancy.
* Patients with tobacco addiction.
* A body mass index (BMI) ≥ 30 before the pregnancy.
* Multiple pregnancies
* A gap of less than 4 weeks between the date of the ultrasound and the date of delivery.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any pregnant patient with a normally progressing pregnancy and reporting for a prenatal screening ultrasound between 31 and 34 weeks amenorrhea.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
fetal growth | at birth
  . During routine prenatal third trimester ultrasonography patients had a fetal weight estimation and measurement of the umbilical resistance index. After delivery we took note of the weight at birth, the term of the delivery, and the time interval between the ultrasound and the delivery, and then we calculated the weight gain on a weekly basis.

REFERENCES:
- [Background] Bolz N, Kalache KD, Proquitte H, Slowinski T, Hartung JP, Henrich W, Bamberg C. Value of Doppler sonography near term: can umbilical and uterine artery indices in low-risk pregnancies predict perinatal outcome? J Perinat Med. 2013 Mar;41(2):165-70. doi: 10.1515/jpm-2012-0042. PMID 23096449
- [Background] Salavati N, Sovio U, Mayo RP, Charnock-Jones DS, Smith GC. The relationship between human placental morphometry and ultrasonic measurements of utero-placental blood flow and fetal growth. Placenta. 2016 Feb;38:41-8. doi: 10.1016/j.placenta.2015.12.003. Epub 2015 Dec 12. PMID 26907381